CLINICAL TRIAL: NCT04797182
Title: Avatrombopag for the Primary Prevention of Thrombocytopenia Induced by Cytarabine-based Chemotherapy in Patients With Lymphoma: An Open, Single-center, Phase II Randomized Controlled Clinical Study
Brief Title: Avatrombopag for the Primary Prevention of Thrombocytopenia Induced by Cytarabine-based Chemotherapy in Patients With Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B2021-034
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Thrombocytopenia; Cytarabine Causing Adverse Effects in Therapeutic Use; Lymphoma
MeSH Terms: conditions — Thrombocytopenia; Lymphoma | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blank control (Experimental): No intervention aiming at preventing thrombocytopenia will be taken after first cycle. Avatrombopag as salvage treatment will be administered to patients suffering from thrombocytopenia with nadir platelet count < 50 × 109/L at a dose of 60mg/day until there is drug-withdrawal indication.
  Interventions: Drug: avatrombopag
- primary prevention (Experimental): As the primary prevention of thrombocytopenia induced by cytarabine-based chemotherapy, Avatrombopag will be administered at a dose of 60mg/day on days -3~-1 and 3~9, for a total of 10 doses. On the condition that patients have platelet counts <50 × 10 9 /L before next cycle, Avatrombopag will be administered at a dose of 60mg/day until there is drug-withdrawal indications. Platelet transfusions were administered to patients when the platelet count was less than 10×109 /L.
  Drug-withdrawal indications:
  PLT ≥ 100×109/L during salvage treatment or platelet count increases by 50×109/L, comparing with baseline level.
  When platelet count is higher than 400×109/L during this study, researchers determine whether avatrombopag is discontinued
  Interventions: Drug: avatrombopag

INTERVENTIONS:
Drug: avatrombopag — avatrombopag,60 mg/d,po

SUMMARY:
This phase 2 trial studies the efficacy and safety of Avatrombopag for the primary prevention of thrombocytopenia induced by cytarabine-based chemotherapy in patients with lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed lymphoma;
* Patients are scheduled to receive cytarabine-based chemotherapy including Ara-C at dose of 4g/m2.
* Eastern Cooperative Oncology Group (ECOG) of 0-1;
* Proper functioning of the major organs: 1) The absolute value of neutrophils (>1.5×10^9/L); platelet count (> 100×10^9/L); Hemoglobin (> 90 g/L); 2) Serum total bilirubin < 1.5 times ULN; Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) < 3 times ULN;3) Serum creatinine <1.5 times Upper Limit Normal (ULN) ; 4) Coagulation function: International Normalized Ratio (INR), Prothrombin Time (PT)< 1.5 times ULN
* Able to use oral drugs
* Patients volunteer to sign an informed consent
* Life expectancy > 3 months;
* Contraceptives are used

Exclusion Criteria:

* Thrombocytopenia unrelated to chemotherapy during six months before screening, including but not limited to hypersplenism, infection and hemorrhage.
* In addtion to CIT caused by lymphoma and chemotherapy,patients also suffer from other blood diseases including ALL, AML, myeloid neoplasms, MDS, myeloproliferative disorders, MM;
* A thrombosis of a coronary artery or vein developed during three months before screening;
* Haemorrhage with severe clinical symptoms, such as gastrointestinal and cerebral hemorrhage;
* Platelet transfusion during two days before randomization;
* Allergic to avatrombopag;
* Participation in any other research about novel agents or devices;
* Pregnant or breastfeeding women;
* Researchers consider it unsuitable for patients to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of grades III and IV thrombocytopenia | 2 years

SECONDARY OUTCOMES:
The durations of any grade thrombocytopenia and grades II, III and IV thrombocytopenia | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China